CLINICAL TRIAL: NCT01590615
Title: Observational, Post-marketing Renal Safety Surveillance Registry in Subjects With Chronic Hepatitis B (HBV) Infection With Decompensated Liver Disease Receiving Nucleotide/Side Therapy
Brief Title: Registry Study for Patients With Chronic HBV Receiving Nucleotide Therapy
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GX-US-174-0172
Record Dates: First submitted 2012-03-20; First posted 2012-05-03 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis B
Keywords: Hepatitis; Hepatitis B; HBV; OLT; MELD; Renal Safety; Liver Transplant
MeSH Terms: conditions — Hepatitis B; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with chronic HBV infection: Participants with decompensated liver disease due to chronic HBV infection, who are receiving or anticipated to receive anti-HBV nucleoside/nucleotide therapy, will be included in the study.
  Interventions: Drug: Anti-HBV nucleoside/nucleotide therapy

INTERVENTIONS:
Drug: Anti-HBV nucleoside/nucleotide therapy — Subjects with chronic HBV infection and with decompensated liver disease who are receiving or anticipated to receive anti-HBV nucleoside/nucleotide therapy will be identified at centers with liver disease expertise where subjects are monitored on a regular basis.

SUMMARY:
This registry will remain open for approximately 5 years (4 years of enrollment + 1 year of follow up). Subjects will be followed until Orthotopic Liver Transplant (OLT), resolution of liver decompensation, death, or conclusion of the registry.

ELIGIBILITY:
Key Inclusion Criteria:

* Estimated glomerular filtration rate (Cockcroft-Gault method)using actual body weight of ≥ 50 mL/min at time of entry into registry
* Negative serologies for HIV, hepatitis C virus (HCV), and/or hepatitis D virus (HDV)
* No history of solid organ or bone marrow transplant
* Currently receiving or anticipated to receive anti-HBV nucleoside/nucleotide therapy within 6 months of inclusion into registry

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with chronic HBV infection receiving or anticipated to receive anti-HBV nucleoside/nucleotide therapy and with decompensated liver disease at time of consent.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-04-26 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a confirmed increase in serum creatinine from baseline of at least one grade | Baseline to Year 5
  The proportion of participants with a confirmed increase in serum creatinine of at least one grade will be calculated as the number of participants with at least one grade increase in serum creatinine from baseline divided by the total number of subjects enrolled over the 4 years of accrual.

SECONDARY OUTCOMES:
Proportion of participants with a confirmed increase in serum creatinine from baseline of at least one grade evaluated using the competing risk cumulative incidence framework | Baseline to Year 5
Proportion of participants with at least one confirmed estimated glomerular filtration rate (eGFR) below 50 mL/min | Baseline to Year 5
Change in eGFR compared to eGFR at baseline by visit window | Baseline to Year 5
Proportion of participants who received appropriate dosing relative to renal function | Baseline to Year 5
Proportion of participants who discontinued anti-hepatitis B virus (HBV) nucleoside/nucleotide therapy due to a renal related event | Baseline to Year 5
Proportion of participants with at least one change in model for end stage liver disease (MELD) score compared to baseline | Baseline to Year 5
Change in MELD score and liver disease status compared to MELD score at baseline by visit window | Baseline to Year 5
Proportion of participants with at least one plasma HBV DNA < 400 copies/mL (69 IU/mL) | Baseline to Year 5
The median number of renal related adverse events per participant over the evaluation period | Baseline to Year 5
  Renal related adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Preferred Term.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (27):
- United States (23):
  - Cedars-Sinai Medical Center for Liver Diseases and Transplantation, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California at San Francisco Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Jackson Memorial Hospital, Miami, Florida
  - Florida Hospital Transplant, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Saint Louis University Hospital, St Louis, Missouri
  - Alegent Creighton Health, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - The Methodist Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - Toronto Liver Centre, Toronto, Ontario